CLINICAL TRIAL: NCT05465486
Title: NeuroSuitUp: Neurorehabilitation Through Synergistic Man-machine Intrefaces Promoting Dormant Neuroplasticity in Spinal Cord Injury
Brief Title: NeuroSuitUp: Neurorehabilitation Through Synergistic Man-machine Interfaces
Acronym: NeuroSuitUp
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Alkinoos Athanasiou, Dr. PhD, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 249473/2019
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injuries
Keywords: Complete SCI; Chronic SCI; Incomplete SCI; Cervical Spine Injury; Neuroplasticity; Robotics; Wearables
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study (Parallel Assignement)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete injury at cervical spine (Experimental): Patients from Greece, 14 y.o. or oder, suffering from chronic complete injury at the cervical spinal cord level (ASIA Impairment Scale A)
  Interventions: Device: Brain-Computer Interface control of robotic arms with augmented reality; Device: Serious game with augmented reality
- Incomplete Injury at cervical spine (Experimental): Patients from Greece, 14 y.o. or oder, suffering from chronic complete injury at the cervical spinal cord level (ASIA Impairment Scale B, C, D, E)
  Interventions: Device: Brain-Computer Interface control of robotic arms with augmented reality; Device: Serious game with augmented reality
- Healthy participants (Active Comparator): Healthy participants, age and sex matched to the participants in the other two arms
  Interventions: Device: Brain-Computer Interface control of robotic arms with augmented reality; Device: Serious game with augmented reality

INTERVENTIONS:
Device: Brain-Computer Interface control of robotic arms with augmented reality — The participants will be trained to modulate self-paced Visual Motor Imagery (VMI) and Kinesthetic Motor Imagery (KMI) under EEG recording in order to achieve BCI-control of a custom-built bimanual arms robot (MERCURY v2.0). In KMI they will be asked to modulate brain waves in order to learn to control the BCI and in VMI they will additionally be projected a visual cue (representation of the intended movement). BCI will be used to control the arms in physical space as well as in an Augmented Reality Environment. Each participant will take part in 3 sessions
  Device: robotic arms MERCURY v2.0 robotic arms is a non-commercial 6-degree-of-freedom anthropomorphic bimanual robotic arms device that was built and developed by the research team of the Medical Physics & Digital Innovation Lab.
Device: Serious game with augmented reality — The participants will don wearable robotics and use them as input to play a dojo-themed immersive serious game intended at tracking participants movement and presenting them with motor tasks to perform. The game wiil be played in a computer screen, as well as in an Augmented Reality Environment. Each participant will take part in 10 sessions
  Device: Wearable robotics The NeuroSuitUp wearable robotics jacket & gloves are non-commercial wearable devices, equiped with inertial motion units, electromyography and electrical muscle stimulation, built and developed by the Medical Physics & Digital Innovation Lab

SUMMARY:
NeuroSuitUp is a multidisciplinary neurophysiological & neural rehabilitation engineering project, developed by the Lab of Medical Physics & Digital Innovation, School of Medicine, Faculty of Health Science Aristotle University of Thessaloniki and supported by a Neurosurgical Department. This research is co-financed by Greece and the European Union (European Social Fund- ESF) through the Operational Programme "Human Resources Development, Education and Lifelong Learning 2014- 2020" in the context of the project ""NeuroSuitUp"" (MIS 5047840). The website for the project can be accessed at https://imedphys.med.auth.gr/project/neurosuitup .

The investigation's primary objectives include the development, testing and optimization of an intervention based on multiple immersive man-machine interfaces offering rich feedback, that include a) mountable robotic arm controlled with wireless Brain-Computer Interface and b) wearable robotics jacket & gloves in combination with a serious game application and c) augmented reality module for the presentation of the previous two, as well as the development and validation of a self-paced neuro-rehabilitation protocol for patients with Cervical Spinal Cord Injury and the study of cortical activity in chronic spinal cord injury.

DETAILED DESCRIPTION:
NeuroSuitUp project's full title is <Neurorehabilitation through synergistic man-machine intrefaces promoting dormant neuroplasticity in spinal cord injury> . It is a multidisciplinary neurophysiological & neural rehabilitation engineering project project, developed by the Lab of Medical Physics & Digital Innovation, School of Medicine, Faculty of Health Science Aristotle University of Thessaloniki and supported by a Neurosurgical Department. This research is co-financed by Greece and the European Union (European Social Fund- ESF) through the Operational Programme "Human Resources Development, Education and Lifelong Learning 2014- 2020" in the context of the project ""NeuroSuitUp"" (MIS 5047840). The website for the project can be accessed at https://imedphys.med.auth.gr/project/neurosuitup .

The NeuroSuitUp project involves:

* A clinical study for rehabilitation of patients with Cervical Spinal Cord Injury (CSCI), using multiple immersive man-machine interfaces (Brain-Computer Interface (BCI) controlled robotic arms device, Wearable Robotics Jacket & Gloves, Serious Gaming Application, Augmented Reality presentation)
* A secondary off-line neurophysiological analysis of brin cortical activation, connectivity and plasticity as well as muscle electrophysiology in patients with CSCI undergoing motor imagery (MI) and BCI training and assistance through electrical muscle stimulation

Milestones of the study:

* The investigators aim to develop, test and optimize an intervention based on multiple immersive man-machine interfaces
* The investigators aim to develop and validate self-paced neuro-rehabilitation protocols for patients with CSCI.
* The investigators aim to identify and study the neurophysiological functionality and alteration of cortical activity in chronic CSCI.

The sensorimotor networks of Spinal Cord Injury (SCI) patients and healthy individuals share similar connectivity patterns of but new functional interactions have been identified as unique to SCI patient networks and can be attributed to both adaptive and maladaptive organization effects after the injury . The importance of such phenomena both as possible prognostic factors and as contributors to patient rehabilitation remains unspecified as of yet. The exact underlying neurophysiological process and the extent that this is modulated by higher-order interactions is also not fully understood. Far more importantly, it has recently demonstrated for the first time partial neurological recovery in complete SCI patients after 5-10 years from the injury through ground-breaking neuro-rehabilitation protocols, integrated into traditional medical and physiotherapy practice. The investigators used rich visual and tactile feedback, virtual reality environments (VRE), BCI controlled exoskeleton and robotic actuators and furthermore documented plasticity effects at the cortical level.

Residual communication between brain and spinal cord plays an important role in possible neurorehabilitation, as even in complete injuries one fourth of nerve fibers crossing the injury level are functionally intact. As such, retraining CNS circuits and promoting plasticity to restore body functions have been recognized among key principles of spinal cord repair by the US National Institute of Neurological Disorders and Stroke (US NIH/NINDS). Nonetheless, existing literature does not yet portray with precision the pathophysiological process and effect of SCI on CNS and the sensorimotor networks. Studies needed to address this issue (such as our study) should be considered, identifing specific questions to be answered through further investigation: a) how and why reorganization of CNS networks is established, b) how this reorganization evolves in time with respect to the severity and chronicity of the injury, c) when can it be considered an adaptive or maladaptive evolution, and d) how can it be promoted or prevented respectively. The gained insight is expected to hold clinical relevance in preventing maladaptive plasticity after SCI through individualized neuro-rehabilitation, as well as in the design of assistive technologies for SCI patients.

This NeuroSuitUp study is a both a pre-clinical neurophysiological investigation on human SCI patients that aims to advance basic knowledge on SCI sequelae to CNS and also a translational implementation in clinical (rehabilitation) practice.. Our analysis aims to eventually help produce a model of CNS function along different stages of SCI (Acute, Sub-acute, Chronic), during different activity (resting state, simple motor tasks, complex sensorimotor activity), differentiate between Complete and Incomplete Injury and ideally being able to predict Negative outcome versus possible Recovery. The NeuroSuitUp project aims to investigate and promote dormant neuroplasticity after chronic SCI at the cervical spine, a type of injury that causes tetraparesis and tetraplegia. Our protocol will deploy training in brain computer interfaces and robotic arms, virtual environments (brain-controlled virtual arms, avatars and augmented reality wearable robotics with sensors and actuators (gloves & jacket) and rich audio/visual/tactile stimuli along with serious gaming applications to enhance motivation. Visual and kinesthetic sensorimotor brain networks will be also studied using high density electroencephalography in order to demonstrate and monitor CNS plasticity.

ELIGIBILITY:
Inclusion Criteria:

* At least 14 yearss of age
* clinical diagnosis of Spinal Cord Injury (SCI evaluated by ASIA Impairment Scale) OR Healthy participants (age and gender matched to SCI patients)
* Sufficient documentation of the injury in case of patients (neurological examination, MRI scan of the injury level, optional additional CT or x-rays).
* Signed informed consent (patients and healthy individuals).

Exclusion Criteria:

* Other neurological condition that has a possibility to significantly affect the neurological status of the participants (or) the ability to control a BCI (or) the neurophysiological recordings:
* Traumatic brain injury
* Central Nervous System tumors
* Multiple Sclerosis
* Amyotrophic Lateral Sclerosis
* Parkinson's disease
* Refractory Epilepsy
* Participation during the last 3months in an another interventional study, the effects of which could affect this study's observations.
* Other grave medical condition that could affect the participation (or) the safety of the participants:
* Cardiac deficiency
* Pulmonary deficiency
* Hearing and visual impairments that can affect the participant's understanding of the intervention and performance.
* Illegal drug use
* Chronic alcoholism

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BCI control (yes/no) | Immediately after the intervention
  Ability of participants to modulate brainwave activity in order to achieve control of the BCI. BCI control is evaluated as achieved or not (there are cases of BCI-illiteracy when the participants cannot modulate their brainwaves in order to control the BCI).
Serious game performance (in-game scoring system) | Immediately after the intervention
  The ability of participants to control the wearables robotic jacket in order to complete in-game tasks and collect more points. The points will be gather be matching the speed and position of the in-game task instructions while receiving assistance from electrical muscle stimulation. The in-game scoring system uses an accumulative scoring regime according to the correct execution of tasks. There is no upper limit to the score and a higher score means better task execution. Counting starts at 0.

SECONDARY OUTCOMES:
Initial Functional Improvement (Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III) | 3 months after first participant in first session
  Daily functionality as measured by the Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III).
  Score ranges from 0 (min, no functional independence) to 100 (max, fully independent).
Intermediate Functional Improvement (Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III) | 6 months after first participant in first session
  Daily functionality as measured by the Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III).
  Score ranges from 0 (min, no functional independence) to 100 (max, fully independent).
Long-term Functional Improvement (Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III) | One year after first participant in first session
  Daily functionality as measured by the Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III).
  Score ranges from 0 (min, no functional independence) to 100 (max, fully independent).
BCI performance classification accuracy | 6 months after first participation in first session
  Achieved performance on BCI at conclusion of BCI sessions for each participant. Measured by classification accuracy (percentage of voluntary non-erroneous commands to overall number of detected commands)
BCI performance by bit rate | 6 months after first participation in first session
  Achieved performance on BCI at conclusion of BCI sessions for each participant. Measured by bit rate (number of commands per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Panos Bamidis, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Laboratory of Medical Physics and Digital Innovation, AUTH, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Athanasiou A, Mitsopoulos K, Praftsiotis A, Astaras A, Antoniou P, Pandria N, Petronikolou V, Kasimis K, Lyssas G, Terzopoulos N, Fiska V, Kartsidis P, Savvidis T, Arvanitidis A, Chasapis K, Moraitopoulos A, Nizamis K, Kalfas A, Iakovidis P, Apostolou T, Magras I, Bamidis P. Neurorehabilitation Through Synergistic Man-Machine Interfaces Promoting Dormant Neuroplasticity in Spinal Cord Injury: Protocol for a Nonrandomized Controlled Trial. JMIR Res Protoc. 2022 Sep 13;11(9):e41152. doi: 10.2196/41152. PMID 36099009
- See also: Study website — https://imedphys.med.auth.gr/project/neurosuitup